CLINICAL TRIAL: NCT04953169
Title: Examining Health Literacy in Biorepository Consents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment delayed during COVID as primary study halted recruitment. Following this, intervention (informational video) was being utilized outside of protocol intervention (informational video)
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Erin Paquette, Assistant Professor of Pediatrics (Critical Care), Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-1092
Record Dates: First submitted 2020-07-02; First posted 2021-07-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pediatric; Critical Illness; Consent
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Intervention: Study participants will be randomized to one of two forms of consent for participation in a biorepository as part of another study in the PICU. One version of consent will be the standard consent used in the study for which they are eligible. The second version of consent will present the standard consent + a biobanking video. The primary outcome will be to assess enrollment in the biorepository based upon consent version. Because the participants will be randomly assigned to groups and this may impact their behavior regarding enrollment in the biorepository, it is an interventional design.
  Secondary outcomes and factors which may correlate with participation will be assessed using qualitative and quantitative measures through an electronic survey. A survey contains questions that will measure knowledge, comprehension, retention, and evaluation of two modes of information delivery, the video + written consent and written information only.
Who Masked: Participant
Masking Description: Each participant will be randomly be assigned either the video or the written consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Other): The video is information regarding biobanking
  Interventions: Other: Biobank Video
- Non-Video (Other): The non-video group will receive a written informed consent
  Interventions: Other: Non-Video

INTERVENTIONS:
Other: Biobank Video — The video describes the process of biobanking with visuals
  Arms: Video
Other: Non-Video — The non-video group will receive a written informed consent
  Arms: Non-Video

SUMMARY:
Previous research has shown that most parents would allow their child's leftover blood to be included in a de-identified biorepository using opt-out consent in an outpatient setting. In a pilot study to evaluate Pediatric Intensive Care Unit (PICU) parents' preferences and comprehension of a written opt-in consent to include their child's sample in a biorepository, the investigators showed 19% of parents did not agree to participate in the Biobank, more than the 8.7% reported in other settings. Parent comprehension varied. and the investigators also noted differential enrollment by sociodemographic factors. Critically ill children and their parents are vulnerable; seeking consent for non-therapeutic research in critical care requires special consideration. Therefore, the goal of this study is to evaluate whether the addition of a stakeholder influenced (parent, clinical research professionals) video aided consent will improve comprehension and rates of enrollment across diverse groups in this high intensity setting.

DETAILED DESCRIPTION:
Previous research has shown that most parents would allow their child's leftover blood to be included in a de-identified biorepository using opt-out consent in an outpatient setting. In a pilot study to evaluate Pediatric Intensive Care Unit (PICU) parents' preferences and comprehension of a written opt-in consent to include their child's sample in a biorepository, the investigators showed 19% of parents did not agree to participate in the Biobank, more than the 8.7% reported in other settings. Parent comprehension varied. and the investigators also noted differential enrollment by sociodemographic factors. Critically ill children and their parents are vulnerable; seeking consent for non-therapeutic research in critical care requires special consideration. Therefore, the goal of this study is to evaluate whether the addition of a stakeholder influenced (parent, clinical research professionals) video aided consent will improve comprehension and rates of enrollment across diverse groups in this high intensity setting.

Previous research showed that most parents would allow their child's leftover blood to be included in a de-identified biorepository using opt-out consent in an outpatient setting. Critically ill children and their parents are vulnerable; seeking consent for non-therapeutic research in critical care requires special consideration. In a pilot study to evaluate Pediatric Intensive Care Unit (PICU) parents' preferences and comprehension of a written opt-in consent to include their child's sample in a biorepository, the investigators showed 19% of parents did not agree to participate in the Biobank, more than the 8.7% reported in other settings. Parent comprehension varied; in general, parents understood the voluntary nature of participation but had limited knowledge of the purposes, risks, and benefits of biorepository research. The investigators showed in an initial single page opt-in consent low rates of comprehension. The investigators also showed differential enrollment by socioeconomic status factors. The goal of this study is to evaluate whether the addition of a stakeholder influenced (parent, clinical research professionals) video aided consent will improve comprehension and rates of enrollment across diverse groups in a pediatric biorepository. To achieve this goal, the study will occur in two phases: first, the investigators will pilot test a survey with up to 20 participants; based on the results of the pilot the investigators will amend the survey, if and as needed, and then begin a larger enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Parents of patients who are nearing readiness for discharge/clinically stable to participate

Exclusion Criteria:

* Other Languages Except For English and Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Rates of enrollment into a biorepository based on consent type | Admission to Discharge from PICU (anticipated up to 6 months but will vary by participant)
  Number of eligible individuals who enroll between groups that watch a biobanking video and those who only receive written consent documents

SECONDARY OUTCOMES:
Parent Race Questionnaire | Baseline 1 time data at time of enrollment
  Parent self-reported race (US Census Categories)
Child Race Chart Extraction | Baseline 1 time data at time of enrollment
  Child race in electronic medical record
Parent Ethnicity Questionnaire | Baseline 1 time data at time of enrollment
  Parent self-reported ethnicity (US Census Categories)
Child Ethnicity Chart Extraction | Baseline 1 time data at time of enrollment
  Child ethnicity in electronic medical record
Parent age Questionnaire | Baseline 1 time data at time of enrollment
  Parent self-reported age in years
Child age Chart Extraction | Baseline 1 time data at time of enrollment
  Child age in years in electronic medical record
Child gender Chart Extraction | Baseline 1 time data at time of enrollment
  Child gender in electronic medical record
Parent gender Questionnaire | Baseline 1 time data at time of enrollment
  Parent self-reported gender
Parent Education Level Questionnaire | Baseline 1 time data at time of enrollment
  Parent self-reported highest level of education
Parent Primary Language Questionnaire | Baseline 1 time data at time of enrollment
  Parent self-reported language
Health Literacy - Parent Self Report on BRIEF Questionnaire | Baseline 1 time data at the time of enrollment
  Four question item completed by parent self report on a Likert scale of familiarity and comfort with health information and completion of medical forms. Three items are scored as: always/often/sometimes/occasionally/never; the last item is scored as not at all/a little bit/somewhat/quite a bit/extremely. Each category is scored 1-5 (in order of how they are written). Higher scores indicate greater health literacy.
Health Literacy - Flesch Kincaid Reading Level | Baseline 1 time data at the time of enrollment
  Consent form grade reading level
Knowledge about biobanking Questionnaire - Semi Structured Comprehension Interview | 2 times - at enrollment (baseline recall/knowledge) and discharge from PICU (retention), expected up to 1 year
  Six question open ended response assessment about the purpose, procedures, risks, benefits, voluntariness, and ability to withdraw from the biorepository. Answers are scored 0,1,2 based on whether they are incorrect, correct but incomplete, or correct and complete.
Satisfaction with the information provided Questionnaire | Baseline 1 time data at the time of enrollment
  8 item questionnaire regarding their satisfaction with the video, with each question rated strongly agree/agree/neutral/disagree/strongly disagree
Satisfaction with understandability Questionnaire - PEMAT-AV for video recipients | Baseline 1 time data at the time of enrollment
  The Patient Education Materials Assessment Tool-Audiovisual is an Agency for Healthcare Quality and Research tool to judge the understandability of audiovisual materials. Relevant questions from a list of available questions can be asked of individuals reviewing AV materials. Each item is ranked agree (1) /disagree (0)/not applicable. The total number of agree/disagree scores are summed and divided by the number of items completed and then multiplied by 100 to get a percentage score of understandability of the materials.
Satisfaction with understandability Questionnaire - PEMAT-Print for standard consent recipients | Baseline 1 time data at the time of enrollment
  The Patient Education Materials Assessment Tool-Print is an Agency for Healthcare Quality and Research tool to judge the understandability of written materials. Relevant questions from a list of available questions can be asked of individuals reviewing written materials. Each item is ranked agree (1) /disagree (0)/not applicable. The total number of agree/disagree scores are summed and divided by the number of items completed and then multiplied by 100 to get a percentage score of understandability of the materials.
What motivated participation - most important factor from Parent Questionnaire | Baseline 1 time data at the time of enrollment
  Parent selection from pre-determined categories of most important factor motivating research participation
What motivated participation - factors that played a role from parent questionnaire | Baseline 1 time data at the time of enrollment
  Survey respondents complete 11 item questionnaire that ranks factors that played a role in their decision as strongly agree/agree/neutral/disagree/strongly disagree.
Parental Anxiety Questionnaire Abbreviated Parental Stress Scale: PICU (A-PSS PICU): | Baseline 1 time data at the time of enrollment.
  7 item measure that assesses environmental factors in the PICU that can contribute to parent stress. Each item is rated on a scale of not experienced/not stressful/minimally stressful/moderately stressful/extremely stressful.
Parental Trust in the Health System/Research Questionnaire | baseline 1 time data at the time of enrollment
  Seven question measure of trust in their physician related to research. Four questions ask about physician explanation of research, ability to ask questions about research, physician recommendations about research if they feel it will cause harm, and whether physicians have ever given treatment as an experiment without consent rated on a Yes/No/I don't know scale. One question asks about whether physicians will prevent unnecessary risk, rated as protect me from risk/sometimes expose me to risk/I don't know. One question asks about whether people will be used as guinea pigs without consent rated as Not at all likely/somewhat likely/Very likely/I don't know. One question asks about prescribing medications as an experiment without consent with choices Not at all/fairly often/Very Often/I don't know.
Satisfaction with decision regarding biorepository enrollment Questionnaire - Decision Regret Scale | discharge data - 1 time data at the time of PICU discharge, expected up to 1 year
  Parents will complete 5 questions on a scale rated strongly agree, agree, neither agree nor disagree, disagree or strongly disagree for each question. Questions assess whether it was the right decision, whether there is any regret, whether they would make the same choice, whther the choice did harm, and whether the choice was a wise one.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Paquette, MD, JD, MBe, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Once we reach target enrollment, we will analyze the data, and prepare a manuscript for publication and grants; the time frame will be approximately Jan 2022 - June 2022.

REFERENCES:
- [Background] Menon K, Ward R; Canadian Critical Care Trials Group. A study of consent for participation in a non-therapeutic study in the pediatric intensive care population. J Med Ethics. 2014 Feb;40(2):123-6. doi: 10.1136/medethics-2012-101075. Epub 2013 Jan 23. PMID 23345569
- [Background] McGregor TL, Van Driest SL, Brothers KB, Bowton EA, Muglia LJ, Roden DM. Inclusion of pediatric samples in an opt-out biorepository linking DNA to de-identified medical records: pediatric BioVU. Clin Pharmacol Ther. 2013 Feb;93(2):204-11. doi: 10.1038/clpt.2012.230. Epub 2012 Nov 21. PMID 23281421
- [Background] Federal Policy for the Protection of Human Subjects. 45 CFR 46. September 8, 2015 2015;80(173):53933-54061.
- [Background] Carman KL, Heeringa JW, Heil SKR, Garfinkel S, Windham A, Gilmore D, Ginsburg M, Sofaer S, Gold M, Pathak-Sen E.. Public Deliberation To Elicit Input on Health Topics: Findings From a Literature Review. Executive Summary. (Prepared by American Institutes for Research under Contract No. 290-2010-000005). AHRQ Publication No. EHC 13-070-EF-1. Rockville, MD: Agency for Healthcare Research and Quality; February 2013. www.effectivehealthcare.ahrq.gov.
- [Background] Rodriguez-Rey R, Alonso-Tapia J. Development of a screening measure of stress for parents of children hospitalised in a Paediatric Intensive Care Unit. Aust Crit Care. 2016 Aug;29(3):151-7. doi: 10.1016/j.aucc.2015.11.002. Epub 2015 Dec 12. PMID 26692497
- [Background] BRIEF Health Literacy Screen: https://healthliteracy.bu.edu/brief
- [Background] Child and Parent Understanding of Clinical Trials: The Semi-Structured Comprehension Interview; Paquette E.T., Najita J., Morley D., Joffe S.; (2015) AJOB Empirical Bioethics, 6 (2) , pp. 23-32.
- [Background] PEMAT AV: https://www.ahrq.gov/ncepcr/tools/self-mgmt/pemat-av.html
- [Background] PEMAT PRINT: https://www.ahrq.gov/ncepcr/tools/self-mgmt/pemat-p.html
- [Background] Corbie-Smith G, Thomas SB, St George DM. Distrust, race, and research. Arch Intern Med. 2002 Nov 25;162(21):2458-63. doi: 10.1001/archinte.162.21.2458. PMID 12437405